CLINICAL TRIAL: NCT01297270
Title: A Phase III, Randomized, Double Blind and Placebo Controlled Study of Once Daily BI 201335 120 mg for 24 Weeks and BI 201335 240 mg for 12 Weeks in Combination With Pegylated Interferon Alpha and Ribavirin in Treatment Naive Patients With Genotype 1 Chronic Hepatitis C Infection.
Brief Title: Efficacy and Safety of BI 201335 (Faldaprevir) in Combination With Pegylated Interferon-alpha and Ribavirin in Treatment-naïve Genotype 1 Hepatitis C Infected Patients (STARTverso 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1220.47; 2010-021716-42 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Results first posted 2015-09-18 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — faldaprevir

ARMS (4):
- PegIFN/RBV (Active Comparator): 48 weeks
  Interventions: Drug: PegIFN/RBV
- BI 201335 for 24 weeks (Experimental): BI 201 335 QD dosing in combination with IFN/RBV
  Interventions: Drug: PegIFN/RBV; Drug: BI201335
- BI201335 for 12 weeks (Experimental): BI 201335 QD doing in combination with PEFG IFN/RBV
  Interventions: Drug: BI201335; Drug: PegIFN/RBV
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI201335 — QD BI 201335
  Arms: BI201335 for 12 weeks
Drug: PegIFN/RBV
  Arms: BI 201335 for 24 weeks; BI201335 for 12 weeks; PegIFN/RBV
Drug: BI201335 — QD (once daily) BI 201335
  Arms: BI 201335 for 24 weeks
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of this trial is to evaluate the efficacy and safety of two different treatment regimens with BI 201335, both in combination with PegIFN/RBV) as compared to standard of care (SOC) with PegIFN/RBV alone.

ELIGIBILITY:
Inclusion criteria:

1. Chronic hepatitis C infection, diagnosed by positive anti-HCV antibodies and detected HCV RNA at screening in addition to:

   1. positive anti-HCV antibodies or detected HCV RNA at least 6 months prior to screening; or,
   2. liver biopsy consistent with chronic HCV infection.
2. HCV genotype 1 infection confirmed by genotypic testing at screening.
3. Therapy-naïve to interferon, pegylated interferon, ribavirin or any antiviral / immunomodulatory drug for acute or chronic HCV infection.
4. HCV RNA = 1,000 IU/mL at screening
5. Documentation of a liver biopsy within 3 years or fibroscan within 6 months of the screening visit.

   Note: If cirrhosis has been previously demonstrated on a biopsy, then biopsies obtained more than 3 years before enrolment need not be repeated. Biopsies can be waived for patients who would be placed at risk from the procedure. Inability to do a liver biopsy should not exclude patients from a trial.
6. Age 18 to 70 years
7. Female patients:

   (c) with documented hysterectomy, (d) who have had both ovaries removed, (e) with documented tubal ligation, (f) who are post-menopausal with last menstrual period at least 12 months prior to screening, or (g) of childbearing potential with a negative serum pregnancy test at screening and Day 1, that, if sexually active, agree to use one of the appropriate medically accepted methods of birth control from the date of screening until 7 months after the last dose of ribavirin in addition to the consistent and correct use of a condom. Patients must agree not to breast-feed at any time from the date of screening until 7 months after the last dose of ribavirin.

   Medically accepted methods of contraception for females in this trial are ethinyl estradiol-containing contraceptives, diaphragm with spermicide substance and intra-uterine device.

   Male patients:
   1. who are documented to be sterile, or
   2. who are without pregnant female partner(s) and consistently and correctly use a condom while their female partner(s) (if of child-bearing potential) use one of the appropriate medically accepted methods of birth control from the date of screening until 7 months after the last dose of ribavirin. It is in the responsibility of the male patient to ensure that his partner(s) is not pregnant prior to screening into the study or becomes pregnant during the treatment and the observation phase.
8. Signed informed consent form prior to trial participation

Exclusion criteria:

1. HCV infection of mixed genotype (1/2, 1/3, and 1/4) diagnosed by genotypic testing at screening.
2. Evidence of acute or chronic liver disease due to causes other than chronic HCV infection.
3. HIV co-infection.
4. Hepatitis B virus (HBV) infection based on presence of HBs-Ag.
5. Active malignancy, or history of malignancy within the last 5 years prior to screening (with an exception of appropriately treated basal cell carcinoma of the skin or in situ carcinoma of the uterine cervix)
6. Active or, history of alcohol or illicit drug abuse other than cannabis within the past 12 months
7. A condition that is defined as one which in the opinion of investigator may put the patient at risk because of participation in this study, may influence the results of this study, or limit the patient¿s ability to participate in this study.
8. Usage of any investigational drugs within 28 days prior to screening, or planned usage of an investigational drug during the course of this study.
9. Received concomitant systemic antiviral, hematopoietic growth factor, or immunomodulatory treatment within 28 days prior to screening. Patients being treated with oral antivirals such as acyclovir, famciclovir or valacyclovir for recurrent herpes simplex infection; or with oseltamivir or zanamivir for influenza A infection, may be screened.
10. Received silymarin (milk thistle), glycyrrhizin, or Sho-saiko-to (SST) within 28 days prior to screening and throughout the treatment phase.
11. Known hypersensitivity to any ingredient of the study drugs.
12. Alpha fetoprotein value >100 ng/mL at screening; if >20 ng/mL and =100 ng/mL, patients may be included if there is no evidence of liver cancer in an appropriate imaging study (e.g., ultrasound, CT scan, or MRI) within last 6 months prior to randomization (Visit 2).
13. Decompensated liver disease, or history of decompensated liver disease, as defined by the presence of: hepatic encephalopathy, ascites, or esophageal variceal bleeding and/or laboratory results of any of the following:

    1. International normalized ratio (INR) of =1.7
    2. Serum Albumin =3.5 g/dL
    3. Serum total bilirubin =2.0 mg/dL (except when the increase is predominately due to unconjugated bilirubin and related to Gilberts syndrome).
14. Pre-existing psychiatric condition that could interfere with the subject¿s participation in and completion of the study including but not limited to prior suicidal attempt, schizophrenia, major depression syndrome, severe anxiety, severe personality disorder, a period of disability or impairment due to a psychiatric disease within the past 5 years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 658 (Actual)
Dates: Start 2011-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (106):
- United States (78):
  - 1220.47.0004 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1220.47.0045 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1220.47.0050 Boehringer Ingelheim Investigational Site, Dothan, Alabama
  - 1220.47.0061 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1220.47.0091 Boehringer Ingelheim Investigational Site, North Little Rock, Arkansas
  - 1220.47.0008 Boehringer Ingelheim Investigational Site, Bakersfield, California
  - 1220.47.0019 Boehringer Ingelheim Investigational Site, Chula Vista, California
  - 1220.47.0010 Boehringer Ingelheim Investigational Site, Coronado, California
  - 1220.47.0033 Boehringer Ingelheim Investigational Site, La Jolla, California
  - 1220.47.0035 Boehringer Ingelheim Investigational Site, La Mesa, California
  - 1220.47.0011 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1220.47.0014 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1220.47.0100 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1220.47.0018 Boehringer Ingelheim Investigational Site, Oceanside, California
  - 1220.47.0059 Boehringer Ingelheim Investigational Site, Poway, California
  - 1220.47.0024 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1220.47.0037 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1220.47.0031 Boehringer Ingelheim Investigational Site, San Francisco, California
  - 1220.47.0082 Boehringer Ingelheim Investigational Site, Englewood, Colorado
  - 1220.47.0049 Boehringer Ingelheim Investigational Site, New Haven, Connecticut
  - 1220.47.0057 Boehringer Ingelheim Investigational Site, Bradenton, Florida
  - 1220.47.0078 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1220.47.0086 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1220.47.0054 Boehringer Ingelheim Investigational Site, Hialeah, Florida
  - 1220.47.0088 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1220.47.0044 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1220.47.0099 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1220.47.0095 Boehringer Ingelheim Investigational Site, Palm Harbor, Florida
  - 1220.47.0074 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1220.47.0022 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1220.47.0039 Boehringer Ingelheim Investigational Site, Columbus, Georgia
  - 1220.47.0052 Boehringer Ingelheim Investigational Site, Decatur, Georgia
  - 1220.47.0013 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1220.47.0055 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1220.47.0062 Boehringer Ingelheim Investigational Site, Vaiparaiso, Indiana
  - 1220.47.0085 Boehringer Ingelheim Investigational Site, Baton Rouge, Louisiana
  - 1220.47.0087 Boehringer Ingelheim Investigational Site, Baton Rouge, Louisiana
  - 1220.47.0101 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 1220.47.0064 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1220.47.0069 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1220.47.0067 Boehringer Ingelheim Investigational Site, Chevy Chase, Maryland
  - 1220.47.0079 Boehringer Ingelheim Investigational Site, Lutherville, Maryland
  - 1220.47.0027 Boehringer Ingelheim Investigational Site, Framingham, Massachusetts
  - 1220.47.0065 Boehringer Ingelheim Investigational Site, Springfield, Massachusetts
  - 1220.47.0023 Boehringer Ingelheim Investigational Site, Tulepo, Mississippi
  - 1220.47.0046 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 1220.47.0066 Boehringer Ingelheim Investigational Site, Neptune City, New Jersey
  - 1220.47.0083 Boehringer Ingelheim Investigational Site, Brooklyn, New York
  - 1220.47.0003 Boehringer Ingelheim Investigational Site, New York, New York
  - 1220.47.0006 Boehringer Ingelheim Investigational Site, New York, New York
  - 1220.47.0038 Boehringer Ingelheim Investigational Site, New York, New York
  - 1220.47.0090 Boehringer Ingelheim Investigational Site, New York, New York
  - 1220.47.0097 Boehringer Ingelheim Investigational Site, The Bronx, New York
  - 1220.47.0053 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1220.47.0021 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1220.47.0098 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 1220.47.0028 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1220.47.0058 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1220.47.0030 Boehringer Ingelheim Investigational Site, Germantown, Tennessee
  - 1220.47.0072 Boehringer Ingelheim Investigational Site, Jackson, Tennessee
  - 1220.47.0032 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 1220.47.0041 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 1220.47.0063 Boehringer Ingelheim Investigational Site, Arlington, Texas
  - 1220.47.0029 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1220.47.0017 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1220.47.0056 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1220.47.0071 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1220.47.0060 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 1220.47.0081 Boehringer Ingelheim Investigational Site, Forth Worth, Texas
  - 1220.47.0009 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1220.47.0068 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1220.47.0016 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1220.47.0015 Boehringer Ingelheim Investigational Site, Burlington, Vermont
  - 1220.47.0042 Boehringer Ingelheim Investigational Site, Annandale, Virginia
  - 1220.47.0043 Boehringer Ingelheim Investigational Site, Falls Church, Virginia
  - 1220.47.0026 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1220.47.0092 Boehringer Ingelheim Investigational Site, Seattle, Washington
  - 1220.47.0073 Boehringer Ingelheim Investigational Site, Milwaukee, Wisconsin
- Canada (15):
  - 1220.47.1011 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1220.47.1012 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1220.47.1001 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1220.47.1003 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1220.47.1016 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1220.47.1007 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 1220.47.1009 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1220.47.1013 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1220.47.1002 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1220.47.1004 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1220.47.1005 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1220.47.1006 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1220.47.1015 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1220.47.1010 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1220.47.1014 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- 1220.47.0034 Boehringer Ingelheim Investigational Site, San Juan, Puerto Rico
- South Korea (7):
  - 1220.47.8204 Boehringer Ingelheim Investigational Site, Pusan
  - 1220.47.8205 Boehringer Ingelheim Investigational Site, Pusan
  - 1220.47.8203 Boehringer Ingelheim Investigational Site, Seongnam
  - 1220.47.8202 Boehringer Ingelheim Investigational Site, Seoul
  - 1220.47.8206 Boehringer Ingelheim Investigational Site, Seoul
  - 1220.47.8207 Boehringer Ingelheim Investigational Site, Seoul
  - 1220.47.8201 Boehringer Ingelheim Investigational Site, Yangsan
- Taiwan (5):
  - 1220.47.8803 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1220.47.8804 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1220.47.8802 Boehringer Ingelheim Investigational Site, Taichung
  - 1220.47.8801 Boehringer Ingelheim Investigational Site, Taipei
  - 1220.47.8805 Boehringer Ingelheim Investigational Site, Taipei

REFERENCES:
- [Derived] Jensen DM, Asselah T, Dieterich D, Foster GR, Sulkowski MS, Zeuzem S, Mantry P, Yoshida EM, Moreno C, Ouzan D, Wright M, Morano LE, Buynak R, Bourliere M, Hassanein T, Nishiguchi S, Kao JH, Omata M, Paik SW, Wong DK, Tam E, Kaita K, Feinman SV, Stern JO, Scherer J, Quinson AM, Voss F, Gallivan JP, Bocher WO, Ferenci P. Faldaprevir, pegylated interferon, and ribavirin for treatment-naive HCV genotype-1: pooled analysis of two phase 3 trials. Ann Hepatol. 2016 May-Jun;15(3):333-49. doi: 10.5604/16652681.1198803. PMID 27049487

RESULTS

PARTICIPANT FLOW:
Groups:
- Faldaprevir 120mg and PegIFN/RBV: Faldaprevir (BI 201335) 120 mg once daily (oral), for 24 weeks, with Pegylated interferon α-2a (PegIFN/RBV), subcutaneous injection/oral. At week 24, if the patients did not achieve early treatment success (ETS) the patient received an additional 24 weeks of PegIFN/RBV alone.
- Faldaprevir 240mg and PegIFN/RBV: Faldaprevir 240 mg once daily (oral), for 12 weeks, with PegIFN/RBV (subcutaneous injection/oral). Followed by an additional 12 weeks of placebo plus PegIFN/RBV. At week 24, if the patients did not achieve early treatment success (ETS) the patient received an additional 24 weeks of PegIFN/RBV alone.
- Placebo and PegIFN/RBV: Placebo (oral) once daily combined with PegIFN/RBV (subcutaneous injection) for 24 weeks, followed by an additional 24 weeks of PegIFN/RBV (oral) alone.
Period: Overall Study
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Started | 262 | 264 | 132
Completed | 217 | 192 | 103
Not Completed | 45 | 72 | 29
Not completed — Adverse Event | 19 | 32 | 5
Not completed — Lack of Efficacy | 15 | 17 | 15
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Protocol Violation | 0 | 2 | 0
Not completed — Withdrawal by Subject | 7 | 15 | 7
Not completed — Other reason not defined above | 3 | 3 | 1
Not completed — Not treated | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized patients who were dispensed study medication and were documented to have taken at least one dose.
Groups:
- Faldaprevir 120mg and PegIFN/RBV: Faldaprevir 120 mg once daily (oral), for 24 weeks, with Pegylated interferon α-2a (PegIFN/RBV), subcutaneous injection/oral. At week 24, if the patients did not achieve early treatment success (ETS) the patient received an additional 24 weeks of PegIFN/RBV alone.
- Total: Total of all reporting groups
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV | Total
Number analyzed (Participants) | 262 | 263 | 132 | 657
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (10.05) | 50.4 (9.40) | 50.2 (8.78) | 50.3 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 109 | 54 | 268
  Male | 157 | 154 | 78 | 389

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response 12 Weeks Post Treatment (SVR12)
Description: Percentage of participants with sustained virologic response 12 weeks post treatment (SVR12) defined as plasma Hepatitis C virus Ribonucleic acid (HCV RNA) level<25 IU/mL (undetected) 12 weeks after the originally planned treatment duration.
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: Full analysis set (FAS) included all randomized patients who were dispensed study medication and were documented to have taken at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 262 | 263 | 132
percentage of participants | 67.9 [62.3 to 73.6] | 64.3 [58.5 to 70.1] | 47.0 [38.5 to 55.5]
Statistical Analysis 1: Comparison: Faldaprevir 120mg and PegIFN/RBV vs Placebo and PegIFN/RBV; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 20.7, 95% CI 2-sided [10.7 to 30.6] — Estimate adjusted for genotype and race using Koch's method, with continuity correction
Statistical Analysis 2: Comparison: Faldaprevir 240mg and PegIFN/RBV vs Placebo and PegIFN/RBV; Test type: Superiority or Other; p = 0.0007, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 17.4, 95% CI 2-sided [7.3 to 27.4] — Estimate adjusted for genotype and race using Koch's method, with continuity correction

2. Secondary Outcome: Sustained Virologic Response 24 Weeks Post-treatment (SVR24)
Description: Percentage of participants with sustained virologic response 24 weeks post-treatment (SVR24), defined as plasma HCV RNA level < 25 IU/mL (undetected) 24 weeks after the originally planned treatment duration.
  Hepatitis C virus Ribonucleic acid (HCV RNA)
Time Frame: 24 weeks post treatment, up to 72 weeks
Population: Full analysis set (FAS) included all randomized patients who were dispensed study medication and were documented to have taken at least one dose of study medication and had SVR data at week 24.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 262 | 263 | 132
percentage of participants | 67.2 [61.5 to 72.9] | 62.7 [56.9 to 68.6] | 46.2 [37.7 to 54.7]
Statistical Analysis 1: Comparison: Faldaprevir 120mg and PegIFN/RBV vs Placebo and PegIFN/RBV; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 20.7, 95% CI 2-sided [10.7 to 30.6] — Estimate adjusted for genotype and race using Koch's method, with continuity correction
Statistical Analysis 2: Comparison: Faldaprevir 240mg and PegIFN/RBV vs Placebo and PegIFN/RBV; Test type: Superiority or Other; p = 0.0014, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 16.6, 95% CI 2-sided [6.5 to 26.7] — Estimate adjusted for genotype and race using Koch's method, with continuity correction

3. Secondary Outcome: Early Treatment Success (ETS)
Description: Percentage of participants with early treatment success (ETS), defined as a plasma HCV RNA level <25 IU/mL (detected or undetected) at week 4 and HCV RNA <25 IU/mL (undetected) at week 8.
Time Frame: Week 4 and week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 262 | 263 | 132
percentage of participants | 80.2 | 79.1 | 15.9

4. Secondary Outcome: ALT Normalisation: ALT in Normal Range at End of Treatment (EOT) When SVR12=YES
Description: The number of participants with alanine aminotransferase (ALT) in normal range at end of treatment (EOT) when patients have sustained virological response 12 weeks post-treatment. BL = Baseline
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 262 | 263 | 132
participants
  SVR12 = Yes | 178 | 169 | 62
  SVR12 = Yes, BL normal to EOT normal | 50 | 52 | 22
  SVR12 = Yes, BL elevated to EOT normal | 89 | 81 | 35
  SVR12 = Yes, No ALT data available at EoT | 0 | 0 | 0

5. Secondary Outcome: ALT Normalisation: ALT in Normal Range at End of Treatment (EOT) When SVR12= NO
Description: The number of participants with alanine aminotransferase (ALT) in normal range at end of treatment (EOT) when patients do not have sustained virological response 12 weeks post-treatment. BL = Baseline
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 262 | 263 | 132
participants
  SVR12 = No | 84 | 94 | 70
  SVR12 = No, BL normal to EOT normal | 21 | 20 | 15
  SVR12 = No, BL elevated to EOT normal | 33 | 44 | 30
  SVR12 = No, No ALT data available at EoT | 3 | 5 | 1

6. Secondary Outcome: ALT Normalisation: ALT in Normal Range 12 Weeks Post-treatment, When SVR12=YES
Description: The number of participants with alanine aminotransferase (ALT) in normal range 12 weeks post-treatment when patients have sustained virological response 12 weeks post-treatment. BL = Baseline
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 262 | 263 | 132
participants
  SVR12 = Yes | 178 | 169 | 62
  SVR12 = Yes, BL normal to SVR12 normal | 52 | 58 | 23
  SVR12 = Yes, BL elevated to SVR12 normal | 105 | 100 | 37
  SVR12 = Yes, No ALT data available at SVR12 visit | 9 | 3 | 0

7. Secondary Outcome: ALT Normalisation: ALT in Normal Range 12 Weeks Post-treatment, When SVR12=NO
Description: The number of participants with alanine aminotransferase (ALT) in normal range 12 weeks post-treatment when patients do not have sustained virological response 12 weeks post-treatment. BL = Baseline
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 262 | 263 | 132
participants
  SVR12 = No | 84 | 94 | 70
  SVR12 = No, BL normal to SVR12 normal | 12 | 11 | 3
  SVR12 = No, BL elevated to SVR12 normal | 13 | 16 | 2
  SVR12 = No, No ALT data available at SVR12 visit | 23 | 34 | 54

8. Secondary Outcome: AST Normalisation: AST in Normal Range at End of Treatment (EOT) When SVR12=YES
Description: The number of participants with aspartate aminotransferase (AST) in normal range at the end of treatment when patients have sustained virological response 12 weeks post-treatment. BL = Baseline
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 262 | 263 | 132
participants
  SVR12 = Yes | 178 | 169 | 62
  SVR12 = Yes, BL normal to EOT normal | 70 | 78 | 26
  SVR12 = Yes, BL elevated to EOT normal | 65 | 51 | 26
  SVR12 = Yes, No AST data available at EoT | 0 | 0 | 0

9. Secondary Outcome: AST Normalisation: AST in Normal Range at End of Treatment (EOT) When SVR12=NO
Description: The number of participants with aspartate aminotransferase (AST) in normal range at the end of treatment when patients do not have sustained virological response 12 weeks post-treatment. BL = Baseline
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 262 | 263 | 132
participants
  SVR12 = No | 84 | 94 | 70
  SVR12 = No, BL normal to EOT normal | 27 | 24 | 17
  SVR12 = No, BL elevated to EOT normal | 27 | 33 | 26
  SVR12 = No, No AST data available at EoT | 3 | 5 | 1

10. Secondary Outcome: AST Normalisation: AST in Normal Range 12 Weeks Post-treatment, When SVR12=YES
Description: The number of participants with aspartate aminotransferase (AST) in normal range 12 weeks post-treatment when patients have sustained virological response 12 weeks post-treatment. BL = Baseline
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 262 | 263 | 132
participants
  SVR12 = Yes | 178 | 169 | 62
  SVR12 = Yes, BL normal to SVR12 normal | 71 | 84 | 29
  SVR12 = Yes, BL elevated to SVR12 normal | 86 | 71 | 30
  SVR12 = Yes, No AST data available at SVR12 visit | 9 | 3 | 0

11. Secondary Outcome: AST Normalisation: AST in Normal Range 12 Weeks Post-treatment, When SVR12=NO
Description: The number of participants with aspartate aminotransferase (AST) in normal range 12 weeks post-treatment when patients do not have sustained virological response 12 weeks post-treatment. BL = Baseline
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Number analyzed (Participants) | 262 | 263 | 132
participants
  SVR12 = No | 84 | 94 | 70
  SVR12 = No, BL normal to SVR12 normal | 13 | 11 | 3
  SVR12 = No, BL elevated to SVR12 normal | 15 | 12 | 1
  SVR12 = No, No AST data available at SVR12 visit | 23 | 34 | 54

ADVERSE EVENTS:
Time Frame: Up to 4 weeks after treatment discontinuation (Up to 48 weeks treatment)
Description: Adverse events (AEs) that pre-existed prior to randomization but worsened during treatment were also considered treatment emergent. All patients who received at least 1 dose of study drug after randomization [safety set (SAF)] were included in the presentation of AE data.
Arm/Group | Faldaprevir 120mg and PegIFN/RBV | Faldaprevir 240mg and PegIFN/RBV | Placebo and PegIFN/RBV
Serious Adverse Events (participants affected / at risk) | 21/262 | 26/263 | 8/132
Other Adverse Events (participants affected / at risk) | 255/262 | 258/263 | 130/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Faldaprevir 120mg and PegIFN/RBV (N=262) | Faldaprevir 240mg and PegIFN/RBV (N=263) | Placebo and PegIFN/RBV (N=132)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Epidermolysis (Congenital, familial and genetic disorders) | 1 | 0 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 | 0
Malaise (General disorders) | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 2 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Infective chondritis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 1
Vulval abscess (Infections and infestations) | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 2
Drug dependence (Psychiatric disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Personality disorder (Psychiatric disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Faldaprevir 120mg and PegIFN/RBV (N=262) | Faldaprevir 240mg and PegIFN/RBV (N=263) | Placebo and PegIFN/RBV (N=132)
Anaemia (Blood and lymphatic system disorders) | 59 | 55 | 27
Neutropenia (Blood and lymphatic system disorders) | 35 | 24 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 13 | 14 | 11
Ocular icterus (Eye disorders) | 3 | 14 | 1
Abdominal pain (Gastrointestinal disorders) | 20 | 23 | 10
Abdominal pain upper (Gastrointestinal disorders) | 15 | 8 | 9
Constipation (Gastrointestinal disorders) | 22 | 14 | 7
Diarrhoea (Gastrointestinal disorders) | 71 | 89 | 23
Dry mouth (Gastrointestinal disorders) | 15 | 16 | 6
Dyspepsia (Gastrointestinal disorders) | 26 | 17 | 3
Nausea (Gastrointestinal disorders) | 99 | 150 | 52
Vomiting (Gastrointestinal disorders) | 40 | 70 | 11
Asthenia (General disorders) | 10 | 19 | 6
Chills (General disorders) | 40 | 38 | 25
Fatigue (General disorders) | 113 | 133 | 70
Influenza like illness (General disorders) | 25 | 14 | 15
Injection site erythema (General disorders) | 13 | 13 | 11
Injection site reaction (General disorders) | 26 | 13 | 4
Pain (General disorders) | 15 | 22 | 9
Pyrexia (General disorders) | 38 | 41 | 20
Hyperbilirubinaemia (Hepatobiliary disorders) | 8 | 25 | 0
Jaundice (Hepatobiliary disorders) | 6 | 24 | 0
Bronchitis (Infections and infestations) | 5 | 14 | 2
Upper respiratory tract infection (Infections and infestations) | 18 | 19 | 9
Weight decreased (Investigations) | 15 | 20 | 10
Decreased appetite (Metabolism and nutrition disorders) | 54 | 63 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 | 36 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 16 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 8 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 47 | 53 | 37
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 12 | 8
Disturbance in attention (Nervous system disorders) | 9 | 14 | 8
Dizziness (Nervous system disorders) | 41 | 39 | 25
Dysgeusia (Nervous system disorders) | 16 | 15 | 3
Headache (Nervous system disorders) | 84 | 81 | 45
Hypoaesthesia (Nervous system disorders) | 8 | 5 | 7
Anxiety (Psychiatric disorders) | 15 | 25 | 14
Depression (Psychiatric disorders) | 32 | 36 | 11
Insomnia (Psychiatric disorders) | 71 | 66 | 38
Irritability (Psychiatric disorders) | 35 | 32 | 27
Chromaturia (Renal and urinary disorders) | 5 | 20 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 46 | 43 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 | 22 | 20
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 12 | 17 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 | 13 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 45 | 51 | 22
Dry skin (Skin and subcutaneous tissue disorders) | 30 | 37 | 15
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 4 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 70 | 94 | 37
Rash (Skin and subcutaneous tissue disorders) | 93 | 105 | 41
Rash macular (Skin and subcutaneous tissue disorders) | 5 | 14 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.